CLINICAL TRIAL: NCT02661438
Title: Multicenter Summative Usability Study of Ciprofloxacin Dry Powder for Inhalation in Subjects With Non-Cystic Fibrosis Bronchiectasis (NCFB) or Chronic Obstructive Pulmonary Disease (COPD) Using Matching Placebo
Brief Title: Summative Usability Study of Ciprofloxacin Dry Powder for Inhalation Using Placebo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 18253
Record Dates: First submitted 2015-12-30; First posted 2016-01-22 (Estimated); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Bronchiectasis; Pulmonary Disease, Chronic Obstructive
Keywords: Usability Test
MeSH Terms: conditions — Bronchiectasis; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Placebo to Ciprofloxacin DPI (Other): Placebo to Ciprofloxacin DPI, 3 doses during test session, 1 additional dose for patients during device training
  Interventions: Drug: Placebo to Ciprofloxacin DPI (BAYQ3939)

INTERVENTIONS:
Drug: Placebo to Ciprofloxacin DPI (BAYQ3939) — Placebo to Ciprofloxacin DPI, 3 doses during test session, 1 additional dose for patients during device training

SUMMARY:
The rationale of this study is to conduct a summative (i.e., validation) usability test of Ciprofloxacin Dry Powder for Inhalation (DPI) and the associated Instructions for Use.

ELIGIBILITY:
Inclusion Criteria

* Subjects (male and female) with non-cystic fibrosis bronchiectasis (NCFB) or chronic obstructive pulmonary disease (COPD)
* Subjects must be aged ≥40
* Subject must be able to independently manage and administer their NCFB/COPD medications

Exclusion Criteria:

* Subjects with recent exacerbation
* Subjects with recent significant hemoptysis in the four weeks before screening (and/or during the screening period)
* Subjects allergic to quinine
* Known chronic bronchial asthma

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2016-01-12 (Actual); Primary Completion 2016-03-17 (Actual); Study Completion 2016-03-17 (Actual)

PRIMARY OUTCOMES:
The user performed the inhalation task based on the given instructions properly (Yes/No). | 1 Day
  The performance was assessed by a test administrator.
The user performed the inhalation task safely (Yes/No). | 1 Day
  The user safety was assessed by a test administrator.
DPI (Dry powder for inhalation) device malfunction (Yes/No). | 1 Day
  The function was assessed by a test administrator.
Subject's subjective feedback (paraphrased) on use-safety and usability | 1 Day

SECONDARY OUTCOMES:
Inhalation time | 1 Day
  Inhalation time is assessed with a stop watch.
User friendliness | 1 Day
  User friendliness is assessd by a questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (2):
- United States (2):
  - Vero Beach, Florida
  - Jamaica, New York